CLINICAL TRIAL: NCT03410251
Title: Long- Term Follow-up of Extraction Socket Management : Clinical Outcomes and Hard Tissue Changes
Brief Title: Long- Term Follow-up of Extraction Socket Management
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Clinical Professor, University of Liege
Other Study IDs: H2016-2 ExMA5
Record Dates: First submitted 2017-07-26; First posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Socket preservation — Teeth were extracted atraumatically and without flap release in patients who have received prophylactic antibiotherapy and local anaesthesia. After checking the integrity of the buccal and palatal bone plate, biomaterial (Bio-Oss®) was introduced into the socket. A connective tissue graft harvested from the palate was inserted and sutured in buccal and palatal pouches in order to cover the socket.
  chlorhexidine spray (0.12%) twice a day and Ibuprofen 600 mg three times/ day were prescribed whereas antibiotics were continued for 5 days. Tooth brushing was banned at the extraction site for 10 days and sutures were removed 10 days after surgery.

SUMMARY:
Twenty-nine patients needing single tooth replacement in aesthetic area were treated by extraction and socket preservation with saddle connective tissue graft between September 2009 and February 2012. Computed Tomography scan were taken at baseline just after the surgery and 3 months later. Long- term evaluation of this particular socket management procedure was evaluated by recalling successfully seventeen of theses patients in June 2016. At this time, a clinical and radiographical consultation was done and Cone Beam CT was taken. Horizontal and vertical bone dimensional changes were then assessed thanks to 3D imaging analysis and esthetic and implants outcomes were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Good general health (ASA 1, 2)
* Controlled periodontitis
* >18 years of age or signed consent by the parents
* Smoking history of<10 cigarettes per day
* Signed informed consent.

Exclusion Criteria:

* Pregnancy or lactation
* Concurrent participation in another trial
* Bone disease or the use of medications that interfered with bone metabolism
* History of head and neck radio- therapy
* Presence of dehiscence or fenestration on bone wall of the socket.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from the Department of Periodontology and Oral Surgery of the University of Liège, Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline Alveolar bone remodeling to 3 months and 6 year: horizontal measurements (based on CBCT, in mm) | Baseline, 3 months, 6 years
  The measurement were done by matching and superimposing CT scans using a three dimensional reconstruction software. Palatal horizontal measurements were calculated by subtracting the buccal horizontal measurements from the total horizontal measurements.
Changes from Baseline Alveolar bone remodeling to 3 months and 6 year : vertical measurements (based on CBCT, in mm) | Baseline, 3 months, 6 years
  The measurement were done by matching and superimposing CT scans using a three dimensional reconstruction software. One vertical measurement was taken on the buccal side, in parallel to the vertical reference line at mid distance between the buccal wall and reference line.

SECONDARY OUTCOMES:
Esthetic outcomes (PES questionnaire) | Approximatively 6 years
  At the cross- sectional long- term evaluation, to analyse the esthetic outcomes of the surgical procedure, the pink esthetic score (PES) was assessed (Fürhauser et al. 2005)
Esthetic outcomes (VAS questionnaire) | Approximatively 6 years
  A VAS questionnaire was given to the patients in order to collect their opinion about the esthetic results.
Implant survival rate (based on criteria of Buser et al., 1990) | Approximatively 6 years
  Success was defined according to the criteria of Buser et al., 1990 which are 1. absence of suppuration (recurring peri implant infection) 2. absence of persistent complaints like pain, foreign body sensation and/or dysesthesia 3. absence of continuous radioluncency area around the implant 4. absence of implant mobility.
Peri-implant bone levels (based on periapical radiography, in mm) | Approximatively 6 years
  The peri- implant bone levels were assessed on periapical radiography using the parallell technique: the distance between the implant shoulder and the first bone to implant contact (DIB) was measured at the mesial and distal aspects using the specific software Image J64 (National Institutes of Health, Bethesda, MD, USA).